CLINICAL TRIAL: NCT01426698
Title: 18 Month Follow Up of Preterm Infants Enrolled in the Cord Clamping Study
Acronym: 18mo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Judith S Mercer, Clinical Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Mercer - 9625
Record Dates: First submitted 2011-08-19; First posted 2011-08-31 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Developmental Delay
Keywords: delayed cord clamping; developmental delay
MeSH Terms: conditions — Learning Disabilities | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate cord clamping (Active Comparator): Infants in this arm will have had immediate cord clamping at birth which is routine care at the hospital
  Interventions: Procedure: delayed cord clamping
- Delayed Cord Clamping (Experimental): Intervention: Following the delivery of the infant, the obstetrician holds the infant approximately 10-15 inches below the mother's introitus at vaginal delivery or 10 to 15 inches below the level of the placenta at Cesarean section. The research nurse records the time when the infant's buttocks are delivered from the vagina or the uterus and counts out the time elapsed in ten second intervals to the obstetrician while he/she is doing the suctioning and drying maneuvers. At 30 to 45 seconds, the obstetrician milks the umbilical cord once, clamps, and cuts it. If the baby appears jeopardized in any way, the obstetrician can alter the protocol for the safety of the infant.
  Interventions: Procedure: delayed cord clamping

INTERVENTIONS:
Procedure: delayed cord clamping — at birth, the obstetrical provider delays the cord clamping for 45 seconds while lowering the infant. At 45 seconds the cord is milked once and then clamped and cut.
  Other Names: DCC

SUMMARY:
The purpose of this study is to examine differences in the long-term effects of immediate versus delayed cord clamping at birth on developmental outcomes of our study infants at 18-22 months corrected age.

DETAILED DESCRIPTION:
The current obstetrical practice at birth in the United States is that the umbilical cord of the very low birth weight (VLBW) infant is clamped immediately. When immediate cord clamping occurs, up to 50% of the fetal-placental blood volume may be left in the placenta acutely increasing vulnerability to hypovolemia (low blood volume). In the investigators previous randomized control trial, it was found that infants who received a simple delay in umbilical cord clamping for 30-45 seconds experienced significantly lower incidence of bleeding in the brain and fewer systemic infections throughout the Neonatal Intensive Care Unit (NICU) stay and had higher scores on muscular control and function at 7 months corrected age. In the investigators current Phase 2 randomized controlled trial, examines the motor functioning of infants randomized to immediate cord clamping (ICC) or delayed cord clamping (DCC) at 7 months corrected age (age based on due date and not the pre-term birth rate).

Our objective for this new grant from the Thrasher Foundation is to examine the differences in the long-term effects of ICC vs. DCC on developmental outcomes of our study infants at 18-22 months corrected age. The investigators hypothesis is that the positive effects of DCC, less bleeding in the brain and less infection, may also result in better motor and mental functioning at 18-22 months corrected age. Differentiation between cognitive and motor function is more obvious in the developing toddler than in younger infants. The diagnosis of cerebral palsy becomes more definitive with age and cognitive skills such as expressive and receptive language continue to emerge.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy between 24 and 31.6 weeks
* singleton fetus
* threatened preterm birth.

Exclusion Criteria:

* Fetuses: congenital anomalies
* Mothers: severe or multiple maternal illnesses
* Drug users or institutionalized or psychotic women

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Motor function | 18-22 months
  Very low birth weight infants in the delayed cord-clamping group will have better motor function at 18-22 months corrected age when compared with VLBW infants in the ICC group.

SECONDARY OUTCOMES:
Mental Functioning | 18 to 22 months
  Very low birth weight infants in the delayed cord-clamping group will have better mental functions at 18-22 months corrected age when compared with VLBW infants in the ICC group.

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Mercer, PhD, CNM, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

REFERENCES:
- [Background] Mercer JS, Vohr BR, Erickson-Owens DA, Padbury JF, Oh W. Seven-month developmental outcomes of very low birth weight infants enrolled in a randomized controlled trial of delayed versus immediate cord clamping. J Perinatol. 2010 Jan;30(1):11-6. doi: 10.1038/jp.2009.170. Epub 2009 Oct 22. PMID 19847185
- [Derived] Wang M, Mercer JS, Padbury JF. Delayed Cord Clamping in Infants with Suspected Intrauterine Growth Restriction. J Pediatr. 2018 Oct;201:264-268. doi: 10.1016/j.jpeds.2018.05.028. Epub 2018 Jun 25. PMID 29954605
- [Derived] Mercer JS, Erickson-Owens DA, Vohr BR, Tucker RJ, Parker AB, Oh W, Padbury JF. Effects of Placental Transfusion on Neonatal and 18 Month Outcomes in Preterm Infants: A Randomized Controlled Trial. J Pediatr. 2016 Jan;168:50-55.e1. doi: 10.1016/j.jpeds.2015.09.068. Epub 2015 Nov 4. PMID 26547399